CLINICAL TRIAL: NCT01144234
Title: Facility-based Intervention to Increase Male Involvement in Antenatal Care and the Prevention Programme of Mother-to-child Transmission of HIV in Eastern Uganda
Brief Title: Male Involvement in Antenatal Care and the Prevention Programme of Mother-to-child Transmission of HIV in Uganda
Acronym: InvolvMaleUg
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre For International Health (Other)
Collaborators: Makerere University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: InvolvMaleUg
Record Dates: First submitted 2010-06-14; First posted 2010-06-15 (Estimated); Last update posted 2013-01-15 (Estimated); Status verified 2013-01

CONDITIONS: HIV Infection
Keywords: Prevention of mother-to-child transmission of HIV-1
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Invitation letter to male spouse (Experimental): In this arm the pregnant women got an invitation letter for the spouse to attend at the next antenatal visit
  Interventions: Behavioral: Invitation letter for male spouse
- Information letter (Placebo Comparator): In this arm the pregnant women got an information letter about antenatal care.
  Interventions: Behavioral: Information letter

INTERVENTIONS:
Behavioral: Invitation letter for male spouse — In this arm the pregnant women got an invitation letter for the spouse to attend at the next antenatal visit
  Arms: Invitation letter to male spouse
Behavioral: Information letter — In this arm the pregnant women got an information letter
  Arms: Information letter

SUMMARY:
HIV /AIDS is a major public health problem in Uganda. The prevention of mother to child transmission of HIV/ AIDS (PMTCT) was launched in Uganda in November 2001 and in Mbale Hospital in May 2002. Currently, PMTCT services have been integrated into mainstream antenatal care services throughout the country.

Though engaging men as partners is a critical component in the PMTCT programme, their involvement has been low. Measures to increase male partner involvement in the PMTCT programmes have not been explored in Uganda.

Objectives: To determine the effect of a written invitation letter to the spouses of women, attending their first antenatal visit on: (a) couple attendance at subsequent antenatal clinic visits; and (b) couple acceptance of HIV testing.

Study site: The study will be carried out at Mbale Regional Referral Hospital in eastern Uganda

Study design: A randomised clinical trial among 1060 (530 intervention and 530 control) new antenatal attendees. The intervention will be a written invitation letter to their spouses.

Outcome measures: The main outcome measure is the proportion of pregnant women who come with their partners for ANC at the subsequent antenatal visit.

Utility: The results of this study will be utilised in re-orienting the ANC services to encourage male participation and hopefully improve the uptake of the PMTCT services at Mbale Regional Referral Hospital.

ELIGIBILITY:
Inclusion Criteria:

* New antenatal mothers (attendees) at Mbale regional referral hospital
* Acceptance to attend at least two subsequent antenatal visits at Mbale hospital

Exclusion Criteria:

* Women attending with their spouses at the first ANC visit
* Refusal to take the letter to her spouse
* Women with inaccessible spouses

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1060 (Actual)
Dates: Start 2010-06; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
proportion of pregnant women who come with their partners | follow-up visit 4 weeks later
  The proportion of pregnant women who come with their partners for antenatal care at the subsequent antenatal visit.

CONTACTS AND LOCATIONS:
Overall Officials: James K Tumwine, MD, PhD, Study Chair — Makerere University; Thorkild Tylleskar, MD, PhD, Study Chair — Centre for International Health, University of Bergen
Locations (1):
- Mbale Regional Referral Hospital, Mbale, Eastern Region, Uganda

REFERENCES:
- [Result] Byamugisha R, Astrom AN, Ndeezi G, Karamagi CA, Tylleskar T, Tumwine JK. Male partner antenatal attendance and HIV testing in eastern Uganda: a randomized facility-based intervention trial. J Int AIDS Soc. 2011 Sep 13;14:43. doi: 10.1186/1758-2652-14-43. PMID 21914207
- [Result] Byamugisha R, Tumwine JK, Semiyaga N, Tylleskar T. Determinants of male involvement in the prevention of mother-to-child transmission of HIV programme in Eastern Uganda: a cross-sectional survey. Reprod Health. 2010 Jun 23;7:12. doi: 10.1186/1742-4755-7-12. PMID 20573250